CLINICAL TRIAL: NCT01324622
Title: Comparison of Cervical Laminectomy to Cervical Laminoplasty* in Patients With Cervical Myelopathy or Myeloradiculopathy Due to Multiple Level Cervical Spinal Canal Stenosis * ARCH™ Fixation System by SYNTHES
Brief Title: Comparison of Cervical Laminectomy to Laminoplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: terminated due to failure to meet enrolment goals
Sponsor: Synthes USA HQ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2442
Record Dates: First submitted 2011-03-23; First posted 2011-03-29 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-10

CONDITIONS: Spinal Cord Diseases
Keywords: Spinal Cord Diseases; Myelopathy; Myeloradiculopathy; Laminectomy; Laminoplasty
MeSH Terms: conditions — Spinal Cord Diseases | interventions — Laminoplasty; Laminectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laminectomy (Active Comparator): Control
  Interventions: Procedure: laminectomy
- Laminoplasty (Active Comparator): Treatment group
  Interventions: Device: Laminoplasty

INTERVENTIONS:
Device: Laminoplasty — Utilizing the ARCH Fixation System (Study device)
  Other Names: ARCH Fixation System
  Arms: Laminoplasty
Procedure: laminectomy — standard procedure
  Arms: Laminectomy

SUMMARY:
The objective of this study is to compare the clinical and radiographic outcomes of multi-level laminectomy to multi-level laminoplasty in the treatment of patients with cervical myelopathy or myeloradiculopathy. The hypothesis for the study is that the laminoplasty group is not inferior to the laminectomy group.

DETAILED DESCRIPTION:
Historically, cervical laminectomy has been proven to be effective in the treatment of symptomatic patients with cervical myelopathy. This standard procedure is employed to accomplish posterior decompression of the cervical spinal cord in patients with multi-level cervical spinal stenosis who have normal or near normal cervical spinal curvature and alignment without associated instability. Laminoplasty was developed in Japan as an alternative to the laminectomy procedure with the intent to reduce post-operative morbidity after dorsal cervical spinal cord decompression, neck pain and to maintain the relative stability of the cervical spine after multi-level decompression.

The goal of both the laminoplasty and laminectomy procedures is to provide spinal cord decompression by enlargement of the spinal canal. A potential benefit of laminoplasty compared to laminectomy is to preserve stability and range of motion of the cervical spine without complete disruption/removal of the posterior laminae, spinous processes and interspinous ligamentous structures. Various authors have described different laminoplasty techniques; all preserve the lamina and expand the size of the spinal canal by fixing the freed or partially freed lamina in a more posterior position.

The primary study hypothesis is that, patients treated with laminoplasty with ARCH fixation (Treatment Group) have clinical and radiographic outcomes as assessed by valid outcomes measures, is not inferior to patients treated with laminectomy (Control Group)

ELIGIBILITY:
Inclusion Criteria: All must be met for inclusion in the study.

* The patient must be at least 18 years of age and have no evidence of developmental anomaly of the cranial cervical junction and/or cervical spine
* The patient has the diagnosis of cervical myelopathy
* The myelopathy or myeloradiculopathy requires a posterior cervical decompression of the spinal canal involving two or more contiguous intervertebral levels including and between C3 and C7
* The patient signs the study informed consent form.

Exclusion Criteria:

* Primary symptoms and signs of cervical radiculopathy (only) without myelopathy.
* Presence of primary focal anterior compression of the cervical spinal cord.
* Ossification of the ligamentum flavum.
* Previous surgery of the cervical spine.
* Tumor, infection, or trauma of the cervical spine or cord.
* Segmental instability - Pregnant or interested in becoming pregnant during the study follow-up period.
* Known sensitivity to device materials.
* Currently being treated or intends to be treated postoperatively with other devices for the same disorder (e.g., electrical stimulation devices, pain control devices, etc.).
* Currently a participant in any other study related to the treatment of cervical spinal disorders.
* Prisoner
* Mentally incompetent, or unable to comply with the follow up regime

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2010-11-01 (Actual); Study Completion 2010-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Lauryssen, MD, Principal Investigator — Tower Orthopaedics; Daniel Riew, MD, Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Tower Orthopaedics, Beverly Hills, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Research Medical Center, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri

REFERENCES:
- [Background] Edwards CC 2nd, Riew KD, Anderson PA, Hilibrand AS, Vaccaro AF. Cervical myelopathy. current diagnostic and treatment strategies. Spine J. 2003 Jan-Feb;3(1):68-81. doi: 10.1016/s1529-9430(02)00566-1. PMID 14589250

RESULTS

PARTICIPANT FLOW:
Groups:
- Laminectomy: Active Comparator: Laminectomy Control, Standard Procedure
- Laminoplasty: Treatment group: Laminoplasty using ARCH Fixation System with allograft bone spacers
Period: Overall Study
Arm/Group | Laminectomy | Laminoplasty
Started | 13 | 11
Completed | 4 | 4
Not Completed | 9 | 7
Not completed — Lost to Follow-up | 7 | 7
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laminectomy | Laminoplasty | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10) | 59 (12) | 58 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24
BMI [Mean (Standard Deviation); unit: kg/m2] | 29 (7) | 30 (4) | 30 (6)

OUTCOME MEASURES:

1. Primary Outcome: Imrovement in Modified Japanese Orthopaedic Assessment (mJOA) Recovery Rate
Description: Number of participants who have mJOA Recovery Rate ≥0%. mJOA Recovery Rate is defined as: mJOA Recovery Rate = ((PostOp Score-PreOp Score)/(17 - Pre-Op Score))*100
Time Frame: 12 months
Population: Number of participants with 12-month follow-up data.
Measure: Number; unit: participants with mJOA Recovery Rate ≥0
Arm/Group | Laminectomy | Laminoplasty
Number analyzed (Participants) | 10 | 10
participants with mJOA Recovery Rate ≥0 | 10 | 10

2. Primary Outcome: Sagittal Angle Success
Description: Success defined as ≤ +15º (kyphosis) as indicated by a neutral lateral radiograph
Time Frame: 12 months
Population: Number of participants with radiographic data available at 12 month visit
Measure: Number; unit: participants with ≤15° sagittal angle
Arm/Group | Laminectomy | Laminoplasty
Number analyzed (Participants) | 8 | 5
participants with ≤15° sagittal angle | 8 | 5

3. Primary Outcome: Incidence of Surgical Interventions
Description: Success defined as a lack of revision, removal or addition of supplemental fixation.
Time Frame: up to 24 months
Measure: Number; unit: participants w/o surgical intervention
Arm/Group | Laminectomy | Laminoplasty
Number analyzed (Participants) | 11 | 13
participants w/o surgical intervention | 10 | 13

4. Secondary Outcome: Pain Scores on the Visual Analog Scale
Time Frame: Up to 24 months
Population: Due to the study's early termination, no data were collected for this outcome.
Units Other Than Participants: Number of patients
Arm/Group | Laminectomy | Laminoplasty
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of patients) | 0 | 0

5. Secondary Outcome: Functional Improvement Using the Neck Disability Index (NDI)
Time Frame: up to 24 months
Population: Due to the study's early termination, no data were collected for this outcome.
Units Other Than Participants: Number of patients
Arm/Group | Laminectomy | Laminoplasty
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of patients) | 0 | 0

6. Secondary Outcome: Quality of Life Improvement Using the SF-12 Scale
Time Frame: up to 24 months
Population: Due to the study's early termination, no data were collected for this outcome.
Units Other Than Participants: Number of patients
Arm/Group | Laminectomy | Laminoplasty
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of patients) | 0 | 0

7. Secondary Outcome: Motor Deficit
Time Frame: up to 24 months
Population: Due to the study's early termination, no data were collected for this outcome.
Units Other Than Participants: Number of patients
Arm/Group | Laminectomy | Laminoplasty
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of patients) | 0 | 0

8. Secondary Outcome: Reflex Evaluation
Time Frame: up to 24 months
Population: Due to the study's early termination, no data were collected for this outcome.
Units Other Than Participants: Number of patients
Arm/Group | Laminectomy | Laminoplasty
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of patients) | 0 | 0

9. Secondary Outcome: Sensory Deficit
Time Frame: up to 24 months
Population: Due to the study's early termination, no data were collected for this outcome.
Units Other Than Participants: Number of patients
Arm/Group | Laminectomy | Laminoplasty
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of patients) | 0 | 0

10. Secondary Outcome: Range of Motion
Time Frame: up to 24 months
Population: Due to the study's early termination, no data were collected for this outcome.
Units Other Than Participants: Number of patients
Arm/Group | Laminectomy | Laminoplasty
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of patients) | 0 | 0

11. Secondary Outcome: Sagittal Canal Diameter
Time Frame: up to 24 months
Population: Due to the study's early termination, no data were collected for this outcome.
Units Other Than Participants: Number of patients
Arm/Group | Laminectomy | Laminoplasty
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of patients) | 0 | 0

12. Secondary Outcome: Extent of Spinal Canal/Cord Decompression
Time Frame: up to 24 months
Population: Due to the study's early termination, no data were collected for this outcome.
Units Other Than Participants: Number of patients
Arm/Group | Laminectomy | Laminoplasty
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of patients) | 0 | 0

ADVERSE EVENTS:
Time Frame: All complications and/or adverse effects were recorded intra-operatively and at each follow-up interval (6 weeks, 6 months, 12 months and 24 months).
Groups:
- Laminectomy: Control laminectomy: standard procedure
- Laminoplasty: Treatment group Laminoplasty: Utilizing the ARCH Fixation System (Study device)
Arm/Group | Laminectomy | Laminoplasty
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/11
Other Adverse Events (participants affected / at risk) | 3/13 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laminectomy (N=13) | Laminoplasty (N=11)
Cervical disc herniation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — As a result of a MVA on 7/31/2009. Subject experienced left arm pain, left foot and leg numbness, intermittent difficulty walking. Diagnosed with C6-C7 herniation with spinal cord compression.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laminectomy (N=13) | Laminoplasty (N=11)
Loss of bladder control (Renal and urinary disorders) | 1 (1) | 0 (0) — Urinary frequency
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness/numbness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Slow enrollment and a low follow-up rate resulted in the early termination of the study and lead to a small numbers of subjects completing the study and limiting the data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less